CLINICAL TRIAL: NCT01505049
Title: Immune Memory After Papillomavirus Vaccination (IMAP-I) Study . DMID 10-0014
Brief Title: Immune Memory After Papillomavirus Vaccination
Acronym: IMAP-1
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Principal Investigator, Mark Mulligan, Professor, Emory University
Other Study IDs: IRB00046117; DMID 10-0014 (Other: Other)
Record Dates: First submitted 2012-01-04; First posted 2012-01-06 (Estimated); Last update posted 2015-07-21 (Estimated); Status verified 2015-07

CONDITIONS: Healthy Volunteers
Keywords: immunology; vaccination; human papillomavirus
MeSH Terms: interventions — Human Papillomavirus Recombinant Vaccine Quadrivalent, Types 6, 11, 16, 18

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — we will retain lymphocyte samples for testing immune function
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (3):
- Previously received all three doses of HPV vaccine: This group will consist of 78 women ages 18 to 30 who have received their third dose of vaccine three or more years ago. Recruitment of this group was completed in Sept 2012.
- Previously received two doses of HPV vaccine: This group will consist of 78 women ages 18 to 30 who have received two doses of the HPV vaccine. The second dose must have been received six or more months ago.
  Interventions: Drug: quadrivalent HPV vaccine
- Unvaccinated Cohort: This group will consist of 45 women who have not received their HPV vaccination. Women ages 18-26 are eligible for this cohort. Recruitment for this group was completed in January 2013.

INTERVENTIONS:
Drug: quadrivalent HPV vaccine — For the group who have received two prior doses of vaccine, the third and final dose of vaccine will be given. For the unvaccinated cohort, women will receive all three doses of the vaccine. The second dose of the vaccine will be given two months after the first dose. The third and final dose of the vaccine will be given six months after the first dose.
  Other Names: Gardasil if the trade name of the quadrivalent HPV vaccine.
  Groups: Previously received two doses of HPV vaccine

SUMMARY:
Vaccines for human papillomavirus (HPV) have been available in the United States since 2006. Early studies have shown a high rate of effectiveness of these vaccines, however it is not known how long this protection will last. The IMAP study will look at various parts of the immune system and potential markers for long lived immune responses to this vaccine.

DETAILED DESCRIPTION:
Three groups of patients will be recruited for this study. One group will be women who have completed all three vaccinations. The second group will be women who are overdue for their final vaccination. We also recruit women who have not been vaccinated previously.

ELIGIBILITY:
Inclusion Criteria:

1. Female ages 18-26 inclusive (18-30 for women who have been previously vaccinated
2. If sexually active and enrolled in unvaccinated group, must use a reliable form of birth control for the first seven months of the study. For the purposes of this protocol a reliable form will be hormonal or barrier contraception. Intrauterine devices and a history of sterilization will also be considered reliable forms of birth control. Abstaining from sex is also a reliable form of contraception.
3. Able to give informed consent
4. Negative urine pregnancy test at enrollment

Exclusion Criteria:

1. Currently pregnant, breast feeding or planning a pregnancy
2. Underlying immunological disease, such as previously diagnosed HIV infection or history of transplantation, history of splenectomy
3. Use of medications with potential immunological effects such as systemic corticosteroids or chemotherapy
4. Prior therapy for cervical dysplasia or cervical cancer such as loop excision, laser ablation, cryotherapy or hysterectomy
5. Unable to comply with protocol
6. Severe allergic reaction (e.g., anaphylaxis) after a previous vaccine dose or to a vaccine component
7. An acute illness, including an oral temperature of 100.4 degrees F within three days of visit

other more specific exclusions may apply to one of the three cohorts

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: we are seeking healthy female volunteers
Sampling Method: Non-Probability Sample
Enrollment: 203 (Actual)
Dates: Start 2012-01; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
To examine markers of immune memory in women receiving quadrivalent HPV vaccine including antibody levels and memory B cells | 2 years after first vaccination

CONTACTS AND LOCATIONS:
Overall Officials: Mark J Mulligan, MD, Principal Investigator — Emory University; Kevin Ault, MD, Principal Investigator — University of Kansas
Locations (1):
- Emory University, Atlanta, Georgia, United States